CLINICAL TRIAL: NCT04461093
Title: Comparison of the Efficacy of Acupressure P6 Point, Dexamethasone and Ondansetron Versus Palonosetron Monotherapy for Preventing Postoperative Nausea and Vomiting in Laparoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mohd Zulfakar Mazlan, MBBS (Other)
Responsible Party: Sponsor-Investigator, Mohd Zulfakar Mazlan, MBBS, Comparison of the efficacy of acupressure P6 point, dexamethasone and ondansetron versus palonosetron monotherapy for preventing postoperative nausea and vomiting in laparoscopic surgery, Universiti Sains Malaysia
Organization: Universiti Sains Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PalanosetronUSM
Record Dates: First submitted 2020-04-15; First posted 2020-07-08 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Palonosetron

STUDY DESIGN:
Intervention Model Description: Double blinded, Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Potential patients are identified and consented for study during pre-operative assessment. Both patients and assessors are blinded in this trial.
  Participants and assessors are being blinded of the treatment or medications given intra-operatively. The acupressure wristband and anti-emetics will be given after general anaesthesia. The wristband will be removed prior to emergence, participants will not aware of the methods used to prevent nausea and vomiting. Postoperative participants will be assessed by independent nurses who are not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Experimental): Group I (n=45)
  1. Acupressure wristband
  2. IV Dexamethasone 8mg
  3. IV Ondansetron 4mg
  Interventions: Other: Acupressure wristband and Palanosetron
- Group II (Active Comparator): Group II (n=45)
  1. IV Palonosetron 0.075mg
  Interventions: Other: Acupressure wristband and Palanosetron

INTERVENTIONS:
Other: Acupressure wristband and Palanosetron — Group 1 Patients with odd numbers labelled form will be Group I patients. They will receive intravenous dexamethasone 8mg during induction. Acupressure P6 wristband is applied after induction and removed prior to emergence to maintain blinding. Intravenous ondansetron 4mg is given prior to skin closure.
  Group 11 Patients with even numbers labelled form will be Group II patients who will receive intravenous palonosetron 0.075mg during induction.

SUMMARY:
Postoperative nausea and vomiting (PONV) is defined as nausea and/or vomiting occurring within 24 hours after surgery, it commonly affects 20-30% patients but as high as 70-80% patients who are deemed high risk for PONV may be affected. PONV may cause unpleasant complications such as dehydration, electrolyte imbalance, suture dehiscence, aspiration of gastric contents, delayed recovery and prolonged hospital stay. Standard guideline recommended combination of anti-emetics to prevent PONV in high risk patients. The commonly used agents are dexamethasone and ondansetron which are cheaper although they are proven to be less effective as single agent when compared with newer agent such as palonosetron. As an adjunct or alternative to pharmacological treatment, acupressure P6 point has gained increasing attention for its possible value in preventing PONV. It is proven that acupressure reduced the incidences of PONV when combined with pharmacological treatment. It is postulated that acupressure active Aβ and Aδ fibres and stimulate the release of β-endorphine from hypothalamus. In addition, it is believed that acupressure might act on dopaminergic, serotonergic and norepinerphrinergic fibres which might has a role in PONV prevention.

DETAILED DESCRIPTION:
This study is designed to compare the efficacy of palonosetron monotherapy versus combination of acupressure P6 point with dexamethasone and ondansetron in preventing PONV. It has been proven that palonosetron is more superior as single agent when compared with acupressure, dexamethasone and ondansetron separately. However, this might not be cost effective as palonosetron is more expensive than the other agents. In addition, the combination therapy has been reported better in preventing PONV when compared with monotherapy. The investigators need to investigate whether the combination of acupressure with dexamethasone and ondansetron exert an effect equal or even better than palonosetron monotherapy. The investigators hypothesis is the combination of acupressure P6 point with dexamethasone and ondansetron provide better prophylaxis againts PONV when compared with palonosetron. The requirement for rescue anti-emetics for combination of acupressure P6 point with dexamethasone and ondansetron group is lesser than palonosetron.

ELIGIBILITY:
Inclusion Criteria:

1. ASA I or II female patients aged 18 - 65 years old in view female patients are at higher risk of postoperative nausea and vomiting.
2. Patients undergoing laparoscopic surgery.
3. High risk for PONV (APFEL score 3-4).

Exclusion Criteria:

1. Patients with known allergic to dexamethasone, ondansetron and wristband.
2. Patients who take anti-emetic, emetogenic drugs and glucocorticoids within 24 hours before surgery.
3. Patients with upper limb disability which affect the application of wristband.
4. Obese patients with BMI > 35 in view acupressure P6 wristband might be too tight to fit patient's wrist which might affect the correct placement of pressure point.
5. Pre-existing vertigo

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative nausea and vomiting immediately, at | Hours 6, postoperative.
The incidence of postoperative nausea and vomiting immediately, at | Hours 12, postoperative
The incidence of postoperative nausea and vomiting immediately, at | Hours 24, postoperative
The incidence of postoperative nausea and vomiting immediately, at | Hours 48, postoperative

SECONDARY OUTCOMES:
The proportion of patients require rescue anti-emetics immediately, | at Hours 6, postoperative.
The proportion of patients require rescue anti-emetics immediately, | Hours 12, postoperative.
The proportion of patients require rescue anti-emetics immediately, | Hours 24, postoperative.
The proportion of patients require rescue anti-emetics immediately, | Hours 48, postoperative.

CONTACTS AND LOCATIONS:
Locations (2):
- Malaysia (2):
  - Mohd Zulfakar Mazlan, MBBS, Kota Bharu, Kelantan
  - Mohd Zulfakar Mazlan, Kota Bharu, Kelantan

IPD SHARING:
Plan to Share IPD: No